CLINICAL TRIAL: NCT00005106
Title: A 96-Week, Randomized, Open-Label, Multicenter Trial to Evaluate the Safety and Tolerability of the Antiretroviral Activity of Stavudine (40mg BID) Plus Lamivudine (150mg BID) Plus Nelfinavir (1250mg BID) Versus Abacavir (300mg BID) Plus Combivir (3TC 150mg/ZDV 300mg BID) Versus Combivir (3TC 150mg/ZDV 300mg BID) Plus Nelfinavir (1250mg BID) in HIV-1 Infected Subjects
Brief Title: A Comparison of Three Anti-HIV Drug Combinations in HIV-Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 264P; ESS40002
Record Dates: First submitted 2000-04-06; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; Stavudine; HIV Protease Inhibitors; Lamivudine; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Adipose Tissue; Lipodystrophy; abacavir
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — lamivudine, zidovudine drug combination; abacavir; Nelfinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to look at the effects of different anti-HIV drug combinations on body fat changes in HIV-positive patients who have never received anti-HIV therapy before.

DETAILED DESCRIPTION:
Patients are randomized to receive stavudine plus lamivudine plus nelfinavir, Combivir (zidovudine plus lamivudine) plus nelfinavir, or Combivir plus abacavir. Patients are stratified into 2 groups based on their screening plasma HIV-1 RNA: (1) greater than 1,000 up to 100,000 copies/ml or (2) greater than 100,000 up to 200,000 copies/ml. Measurements and evaluations for assessment of body fat composition, virologic and immunologic outcomes, markers of alterations in carbohydrate and lipid metabolism, and safety are performed at Baseline, Weeks 4, 8, 16, 24, and every 12 weeks thereafter until Week 96 or withdrawal. In addition, health-related quality of life and health care resource utilization data are collected at specified treatment visits.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Are HIV-positive.
* Have a CD4 count greater than 50 cells/mm3.
* Have a viral load greater than 1,000 copies/ml but less than 200,000 copies/ml.
* Have never received anti-HIV medications before. (However, less than 1 week of therapy with lamivudine or a protease inhibitor and less than 4 weeks of therapy with other nucleoside reverse transcriptase inhibitors [NRTIs] is allowed. No therapy with nonnucleoside reverse transcriptase inhibitors [NNRTIs] is allowed.)
* Cannot bear children or agree to use effective methods of birth control during the study. Hormonal methods of birth control (such as birth control pills) are not considered effective for this study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an active AIDS-defining opportunistic infection or disease that, in the doctor's opinion, would make them unable to participate.
* Are unable, in the opinion of the doctor, to follow the dosing schedule and follow-up visit schedule.
* Have a substance abuse problem that would interfere with taking the medications correctly or attending the clinic visits.
* Are enrolled in another study.
* Cannot take medications by mouth or absorb drugs.
* Have hepatitis.
* Have a serious medical condition such as diabetes, congestive heart failure, or other heart disease.
* Need chemotherapy or radiation therapy (except for local treatment of Kaposi's sarcoma).
* Are taking certain medications.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Clinical Research Ctr Inc, Tucson, Arizona
  - Longbeach Memorial Med Ctr, Longbeach, California
  - Good Samaritan Hosp, Los Angeles, California
  - THE Clinic, Los Angeles, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Maxine Liggins, Los Angeles, California
  - UCLA Care Ctr, Los Angeles, California
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - San Francisco Gen Hosp, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Children's Diagnostic Treatment Ctr, Fort Lauderdale, Florida
  - Community Health Care, Fort Lauderdale, Florida
  - Comprehensive Care Center, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - South Shore Hosp, Miami, Florida
  - Orange County Health Dept, Orlando, Florida
  - Immunity Care and Research Inc, Plantation, Florida
  - Daniel Seekins, Tampa, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Ponce de Leon Ctr, Atlanta, Georgia
  - Philip Brachman, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - HIV Outpatient Clinics / LA State Univ Med Ctr, New Orleans, Louisiana
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - South Jersey Infectious Diseases Inc, Somers Point, New Jersey
  - WNC Community Health Services, Asheville, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Summa Health System, Akron, Ohio
  - MCP Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Miriam Hosp, Providence, Rhode Island
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Thomas Street Clinic, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia